CLINICAL TRIAL: NCT06709937
Title: Prospective Multicenter Registry of Patients With Skin Metastases From Breast Cancer Treated With Electrochemotherapy
Acronym: GISEL
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Corrado Giacomo, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2509
Record Dates: First submitted 2024-11-20; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Electrochemotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with metastatic breast carcinoma: In patients with metastatic breast carcinoma, the skin is affected in 5-30% of cases. Although constituting a relatively rare event in absolute terms, the onset of cutaneous metastases generally represents an unfavorable prognostic factor (due to synchronous progression of disease in other sites), as well as a condition of difficult therapeutic management. Even in the most favorable cases, cutaneous metastases often lead to a deterioration in the quality of life of patients, linked to their psychological impact and associated symptoms. It is crucial that patients receive timely and effective treatment. In these cases, various therapeutic options are discussed by a multidisciplinary team, and the patient is typically evaluated for systemic treatment (chemotherapy, endocrine therapy, targeted therapy).
  Interventions: Other: Prospective multicenter registry of patients with cutaneous metastases from breast carcinoma treated with electrochemotherapy.

INTERVENTIONS:
Other: Prospective multicenter registry of patients with cutaneous metastases from breast carcinoma treated with electrochemotherapy. — electrochemotherapy.

SUMMARY:
Electrochemotherapy (ECT) has been proposed as a new therapeutic option for palliating cutaneous metastases from breast carcinoma.

DETAILED DESCRIPTION:
Electrochemotherapy

Recently, electrochemotherapy (ECT) has been proposed as a new therapeutic option for palliating cutaneous metastases from breast carcinoma. Over the last decade, ECT has represented an innovative and effective local/regional therapy in the field of dermato-oncology. In brief, it consists of combining chemotherapy with the local application (at the tumor site) of electric pulses. Through the application of short and intense electric pulses, a physical phenomenon (reversible electroporation) occurs, consisting of the temporary opening of pores through the cell membrane, increasing its permeability. This mechanism allows for the diffusion of poorly permeable drugs into the cytoplasm. Once the transmembrane pores close, after a few milliseconds, the final effect is the concentration of the chemotherapeutic drug inside the cell and an increase in its cytotoxic effect. The enhancement of cytotoxic action ranges from 80 (in the case of cisplatin) to 8000 times (in the case of bleomycin).

Clinical experience with electrochemotherapy

The initial clinical experiences in treating patients with cutaneous metastases using ECT demonstrated very promising results in tumors of various histotypes. After the standardization of the method, studies published over the last decade provide extensive evidence that ECT has high antitumor activity. The most extensive experience has been primarily gathered in patients with superficial metastases from melanoma and breast carcinoma and has also been the subject of a meta-analysis comparing different "skin-directed" therapies.

In current clinical practice, ECT is employed as a complementary or alternative treatment in the management of tumors and cutaneous metastases that are not surgically resectable or not amenable to treatment with radiotherapy or systemic oncologic therapies. Thanks to its relative ease of application and low toxicity profile, ECT represents an effective tool for palliating symptomatic superficial metastases (bleeding, ulcerated, painful), ensuring preservation of the patient's quality of life regarding aspects related to the presence of the disease at the cutaneous level.

The main advantages of treatment with ECT are represented by the following factors:

* possibility of administration on a day-surgery/day-hospital basis
* preservation of healthy tissues
* use of relatively low-toxicity antitumor drugs
* possibility of repeated treatment
* favorable toxicity profile (side effects are mostly cutaneous)
* good patient compliance

The use of the method has progressively increased, especially in Europe, following the publication of European Standard Operative Procedures of Electrochemotherapy (ESOPE) in 2006. These guidelines served as the basis for conducting a multicenter European study (ESOPE Study) that demonstrated the feasibility of the indicated operative modalities and the safety of the procedure.

Clinical experience with electrochemotherapy in breast carcinoma

Clinical experiences in subsequent years have been summarized in two recent meta-analyses, mainly based on studies in patients with melanoma and breast carcinoma, where ECT demonstrated a complete response rate of 59% and 57.5%, respectively. A phase 2 study conducted at the Veneto Oncology Institute in Padua on 34 patients with recurrent cutaneous lesions on the thoracic wall reported an overall response rate of 87%, with 40% of patients achieving a complete and lasting response on the treated lesions. Comparable results have been obtained in other smaller experiences reported in the literature.

More recently, a multicenter retrospective study was published by the Italian Senological Group for Electrochemotherapy (GISEL) based on 125 patients with cutaneous metastases from breast carcinoma. According to the data from this study, the response rate to ECT was 90%, with 58% of patients reporting a complete response. In this study, tumor size (<3cm), presence of hormonal receptors, low proliferative index (Ki-67), absence of tumor ulceration, and absence of visceral metastases were predictive factors for a complete response to treatment. Based on this data and subdividing patients into intrinsic subtypes indicated by the St. Gallen classification, patients with "luminal A-like" type tumors reported a significantly higher complete response rate than all others (73.9% vs 54.7%, P=0.02).

If these preliminary observations were confirmed by a prospective study on a larger case series, it could improve the criteria for selecting patients with breast carcinoma eligible for ECT treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cutaneous metastases from breast carcinoma not surgically resectable;
* No indications for radiotherapy treatment;
* Patients not eligible or not fully responsive to systemic oncologic treatments;
* Maximum depth of the lesion from the skin surface: 3 cm;
* Patient's life expectancy exceeding 4 months;
* Normal hematologic, hepatic, and renal function;
* Performance status ≤2 according to the ECOG scale.

Exclusion Criteria:

* History of allergic reactions to bleomycin or cisplatin;
* Exceeding the maximum cumulative dose of bleomycin (250,000 IU/m2);
* Peripheral neuropathy (in case of cisplatin use);
* Severe hepatic or renal insufficiency;
* History of epilepsy;
* Presence of a pacemaker;
* Severe cardiac arrhythmias (In patients with a history of cardiac arrhythmia, a cardiological evaluation will be performed, and treatment will be applied in the presence of an anesthesiologist. The presence of any type of pacemaker precludes treatment on the thoracic wall);
* Pregnancy or breastfeeding;
* Unavailability for follow-up visits;
* Altered respiratory function or presence of pulmonary fibrosis.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: To test the hypothesis of a significant difference between two proportions (73.9% vs 54.7%) using a one-tailed likelihood ratio test, with a statistical power of 90% and a target significance level of 5%, 351 patients are required (64 in the "luminal A-like" group and 287 in the non-"luminal A-like" group).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The rate of local response in the entire study population and in the subgroups | 1-3-6 months
  Confirmation with a large case series of the results obtained in the multicenter study by the GISEL group

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Corrado, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy